CLINICAL TRIAL: NCT03171740
Title: Premedication With Intranasal Dexmedetomidine or Midazolam for Prevention of Emergence Agitation in Children: Superiority Randomized Clinical Trial
Brief Title: Premedication With Intranasal Dexmedetomidine or Midazolam for Prevention of Emergence Agitation in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, Head of anesthesiology, Brasilia University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VictorSoutoAnestesiologia2017
Record Dates: First submitted 2017-05-27; First posted 2017-05-31 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Emergence Delirium
Keywords: Emergence Delirium; Emergence Agitation; premedication; dexmedetomidine; midazolam
MeSH Terms: conditions — Emergence Delirium | interventions — Dexmedetomidine; Midazolam; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: All participants will receive an intranasal and an oral drug. One group will receive oral midazolam and intranasal saline, the other will receive oral saline and intranasal dexmededomedine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will not know which group they will be allocated. The anesthesia care provider will not know which premedication the patient received because another professional, who is not from the research team, will provide it to the child. The investigator and outcome assessor will only know the allocated group latter by a code which will be revealed after the end of the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Children will receive 1mcg/kg intranasal dexmedetomidine and oral saline, 30 minutes before going to operation theater.
  Interventions: Drug: Dexmedetomidine; Drug: Oral saline
- Midazolam oral solution (Active Comparator): Children will receive 0,5mg/kg oral midazolam and intranasal saline, 30 minutes before going to operation theater.
  Interventions: Drug: Midazolam oral solution; Drug: Nasal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Intranasal dexmedetomidine, 1mcg/kg (it is a 100mcg/ml solution)
  Other Names: Precedex
  Arms: Dexmedetomidine
Drug: Midazolam oral solution — Oral midazolam, 0.5mg/kg (its a 2mg/ml solution)
  Arms: Midazolam oral solution
Drug: Oral saline — Oral saline, 0.25ml/kg
  Other Names: 0.9% Saline solution
  Arms: Dexmedetomidine
Drug: Nasal saline — Nasal saline 0.01ml/kg
  Other Names: 0.9% Saline solution
  Arms: Midazolam oral solution

SUMMARY:
Study where children will receive one premedication, either intranasal dexmedetomidine or oral midazolam, to reduce agitation on emergence of anesthesia. The hypothesis is that dexmedetomidine is superior but previous studies lack quality.

DETAILED DESCRIPTION:
Children will be randomized to receive, either midazolam (0.5mg/kg) or dexmedetomidine (1mcg/kg), as anesthetic premedication. Emergence agitation will be assessed by PAED scale.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for amygdalectomy
* American Society of Anesthesiologists Physical Status PI or PII
* Absence of congenital neuropathy
* Absence of cardiac pathology (any)
* Intolerance to one of the studied drugs.

Exclusion Criteria:

* Protocol violation
* Need to transfer for ICU intubated

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Emergence agitation | 15 minutes
  Anesthesiologist provider's reported score on PAED (Paediatric Anesthesia Emergence Scale) during the first 15 minutes after the extubation. The PAED consists of four items. Each item is scored 0-4 yielding a total between 0 and 20.

SECONDARY OUTCOMES:
Bradycardia | 2 hours
  It is defined as a heart rate lower than the expected for the age or a drop higher than 30% of the patient's lowest previous heart rate registered. It will be measured using pletysmography and ECG beat-by-beat during the surgery and it will be true if it occurs at least once.
Hypotension | 2 hours
  It is defined as a mean arterial pressure lower than the expected for the age or a drop higher than 30% of the patient's lowest previous mean arterial pressure registered. It will be measured using oscillatory method every 5 minutes during the surgery and it will be true if it occurs at least once.
Intraocular pressure | 15-minutes
  It will be measured in the first 15 minutes after the induction of general anesthesia using an ocular tonometer. It is measured in mmHg.
Respiratory depression | 30 minutes
  Anesthesiologist provider's reported incidence respiratory depression in the child, before induction of general anesthesia. It will be true if the respiratory rate is slow for the age and the variable is dichotomic (true or false).
Paradoxal agitation | 30 minutes
  Anesthesiologist provider's reported incidence paradoxal agitation in the child, before induction of general anesthesia. The assessment subjective and the variable is dichotomic (true or false).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MN Guimarães, MD, Study Chair — University of Brasilia
Locations (1):
- University Hospital of Brasilia University, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Plan to share the database used for analysis, without any variable that may help to identify individuals (such as name, register), to facilitate meta-analysis and re-analysis.